CLINICAL TRIAL: NCT01606254
Title: A Repeated Dose Study of JNS010 (Paliperidone Palmitate) in Patients With Schizophrenia
Brief Title: A Pharmacokinetic and Safety Study of Paliperidone Palmitate (JNS010) in Participants With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013612; PALM-JPN-2 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2012-05-15; First posted 2012-05-25 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Palmitate; JNS010
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paliperidone palmitate 50 mg (Experimental): Paliperidone palmitate 50 milligram (mg) intramuscular (into the muscle) injection on Days 1, 8, 36 and 64.
  Interventions: Drug: Paliperidone palmitate
- Paliperidone palmitate 100 mg (Experimental): Paliperidone palmitate 100 mg intramuscular injection on Days 1, 8, 36 and 64.
  Interventions: Drug: Paliperidone palmitate
- Paliperidone palmitate 150 mg (Experimental): Paliperidone palmitate 150 mg intramuscular injection on Days 1, 8, 36 and 64.
  Interventions: Drug: Paliperidone palmitate
- Paliperidone palmitate 150/ 50 mg (Experimental): Paliperidone palmitate 150 mg intramuscular injection on Day 1 and paliperidone palmitate 50 mg intramuscular injection on Days 8, 36 and 64.
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Paliperidone palmitate aqueous suspension for injection 0.5, 1.0, 1.5 milliliter equivalent to 50, 100, 150 mg paliperidone respectively as intramuscular injection on Days 1, 8, 36 and 64.
  Other Names: JNS010

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) and safety of paliperidone palmitate in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), open-label (all people know the identity of the intervention), randomized (the study drug is assigned by chance), parallel-group (Each group of participants will be treated at the same time), comparison study to assess the pharmacokinetics and safety of paliperidone palmitate (study medication) in participants with schizophrenia. The study comprises a 64-day Treatment period and a 155-day Follow-up period. The participants will be randomly assigned to one of the four study groups. The study medication will be administered on Days 1, 8, 36 and 64. Pharmacokinetics of the study medication will be assessed as primary outcome. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria

* Participants who have been diagnosed with schizophrenia in accordance with the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV)
* Participants may be inpatients or outpatients
* Participants who have been taking an oral antipsychotic medication for at least 28 days before the date of informed consent
* Participants with a Positive and Negative Syndrome Scale (PANSS) score of less than or equal to 4 (moderate) at screening
* Participants who have taken risperidone by the start of investigational treatment and the record can be confirmed Exclusion Criteria
* Participants who have been diagnosed with a mental disease other than schizophrenia in accordance with the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV)
* Participants who have been diagnosed with substance-related disorders (except nicotine and caffeine dependence)
* Participants with complicated parkinson's disease (a progressive disorder of the central nervous system, seen usually in older persons, in which there is muscle weakness, trembling and sweating)
* Participants with a complication of or with a history of convulsive disease such as epilepsy (seizure disorder)
* Participants with a complication of or with a history of cerebro-vascular accident (stroke), neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness) or physical exhaustion associated with the state of dehydration (lose of water and minerals in the body) or malnutrition

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Ichikawa, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Palmitate 50 mg: Paliperidone palmitate (JNS010) 50 milligram (mg) intramuscular (into the muscle) injection administered on Days 1, 8, 36 and 64.
- Paliperidone Palmitate 100 mg: Paliperidone palmitate 100 mg intramuscular injection administered on Days 1, 8, 36 and 64.
- Paliperidone Palmitate 150 mg: Paliperidone palmitate 150 mg intramuscular injections administered on Days 1, 8, 36 and 64.
- Paliperidone Palmitate 150/ 50 mg: Paliperidone palmitate 150 mg intramuscular injection administered on Day 1 and paliperidone palmitate 50 mg intramuscular injection administered on Days 8, 36 and 64.
Period: Overall Study
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Started | 14 | 14 | 14 | 14
Completed | 12 | 10 | 14 | 11
Not Completed | 2 | 4 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone Palmitate 50 mg: Paliperidone palmitate 50 milligram (mg) intramuscular injection administered on Days 1, 8, 36 and 64.
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (13.8) | 45.2 (11.1) | 48.7 (11.8) | 49.4 (12.1) | 47.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 6 | 16
  Male | 12 | 9 | 11 | 8 | 40
Number of Participants with Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score [Number; unit: Participant] — Drug Induced Extra-Pyramidal Symptoms Scale (DIEPSS) is a scale used to evaluate the severity of drug induced extra-pyramidal symptoms occurring during antipsychotic drug treatment. Scale consists of 8 individual symptom scales with scores ranging from 0 (none/normal) to 4 (severe). The total score is the average of the 8 item scores, for a total range of 0 (normal) to 4 (severe). Overall severity was assessed at 5 levels (0 [none, normal]; 1 [Very Mild]; 2 [Mild]; 3 [Moderate]; 4 [severe]).
  Participant
    None | 8 | 8 | 5 | 5 | 26
    Very mild | 6 | 6 | 8 | 9 | 29
    Mild | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Paliperidone Pre-dose Plasma Concentration (Cpredose) at Day 8
Description: The pre-dose plasma concentration (Cpredose) at Day 8 is defined as the plasma concentration obtained before a dose is given on Day 8. The mean Cpredose at Day 8 was measured in nanogram per milliliter (ng/ml).
Time Frame: Day 8
Population: Pharmacokinetic analysis set included all participants who received the study treatment and whose plasma drug concentrations were available. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 14 | 13 | 14
ng/ml | 5.85 (4.47) | 7.28 (4.92) | 28.4 (29.2) | 12.1 (7.46)

2. Primary Outcome: Paliperidone Pre-dose Plasma Concentration (Cpredose) at Day 36
Description: The Cpredose at Day 36 is defined as the plasma concentration obtained before a dose is given on Day 36. The mean Cpredose at Day 36 was measured in ng/ml.
Time Frame: Day 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 12 | 14 | 12
ng/ml | 6.77 (3.75) | 14.5 (5.76) | 23.4 (18.6) | 19.5 (16.1)

3. Primary Outcome: Paliperidone Pre-dose Plasma Concentration (Cpredose) at Day 64
Description: The Cpredose at Day 64 is defined as the plasma paliperidone concentration obtained before a dose is given on Day 64. The mean Cpredose at Day 64 was measured in ng/ml.
Time Frame: Day 64
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
ng/ml | 6.86 (3.31) | 15.1 (9.16) | 22.9 (16.3) | 14.3 (9.01)

4. Primary Outcome: Paliperidone Pre-dose Plasma Concentration (Cpredose) at Day 92
Description: The Cpredose at Day 92 is defined as the plasma paliperidone concentration obtained after the treatment interval of the study drug (that is 4 weeks) passed after the final dose (Day 92). The mean Cpredose at Day 92 was measured in ng/ml.
Time Frame: Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
ng/ml | 8.41 (4.51) | 15.2 (6.21) | 25.4 (16.8) | 13.5 (6.38)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Paliperidone
Description: The Cmax is defined as maximum observed analyte concentration.
Time Frame: Days 1, 8, 15, 22, 36, 50, 64, 67, 71, 74, 78, 85, 92, 106, 120, 134, 162, 190, 218 and early withdrawal
Population: Pharmacokinetic analysis set included all participants who received the study medication and whose plasma drug concentrations were available. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
ng/ml | 13.7 (7.52) | 33.5 (19.8) | 43.1 (30.3) | 21.6 (12.9)

6. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Paliperidone
Description: The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time Frame: Days 1, 8, 15, 22, 36, 50, 64, 67, 71, 74, 78, 85, 92, 106, 120, 134, 162, 190, 218 and early withdrawal
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
Days | 10.99 [1.99 to 21.01] | 7.89 [5.97 to 21.81] | 7.50 [2.93 to 27.01] | 3.82 [0.71 to 7.07]

7. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: The AUCtau is a measure of the plasma paliperidone concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Time Frame: Days 1, 8, 15, 22, 36, 50, 64, 67, 71, 74, 78, 85, 92, 106, 120, 134, 162, 190, 218 and early withdrawal
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
nanogram*hour per milliliter | 7081 (3581) | 15898 (7535) | 21853 (15534) | 11109 (5390)

8. Primary Outcome: Plasma Paliperidone Concentration at Steady State (Css av)
Description: The Css av is defined as value of average analyte concentration at steady-state (after 4 Intramuscular Injections of Paliperidone Palmitate).
Time Frame: Days 1, 8, 15, 22, 36, 50, 64, 67, 71, 74, 78, 85, 92, 106, 120, 134, 162, 190, 218 and early withdrawal
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
ng/ml | 10.7 (5.42) | 23.9 (11.4) | 32.8 (23.1) | 16.7 (8.28)

9. Primary Outcome: Paliperidone Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Days 1, 8, 15, 22, 36, 50, 64, 67, 71, 74, 78, 85, 92, 106, 120, 134, 162, 190, 218 and early withdrawal
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 10 | 10 | 9 | 11
Days | 68.1 (48.0) | 58.5 (29.1) | 95.5 (98.8) | 104.4 (97.1)

10. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 8
Description: The DIEPSS is a scale used to evaluate the severity of drug induced extra-pyramidal symptoms occurring during antipsychotic drug treatment. Scale consists of 8 individual symptom scales with scores ranging from 0 (none/normal) to 4 (severe). The total score is the average of the 8 item scores, for a total range of 0 (normal) to 4 (severe). Overall severity was assessed at 5 levels (0 [none, normal]; 1 [Very Mild]; 2 [Mild]; 3 [Moderate]; 4 [severe]).
Time Frame: Day 8
Population: Safety analysis set included all participants who were enrolled in the study and received the study medication at least once.
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14
Participants
  None | 6 | 9 | 6 | 6
  Very mild | 8 | 5 | 6 | 7
  Mild | 0 | 0 | 2 | 1

11. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 22
Description: as for outcome 10
Time Frame: Day 22
Population: Safety analysis set included all participants who were enrolled in the study and received the study medication at least once. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 13 | 14 | 14
Participants
  None | 7 | 7 | 6 | 6
  Very mild | 7 | 6 | 7 | 8
  Mild | 0 | 0 | 1 | 0

12. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 50
Description: as for outcome 10
Time Frame: Day 50
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 12 | 14 | 12
Participants
  None | 11 | 7 | 8 | 6
  Very mild | 3 | 5 | 5 | 6
  Mild | 0 | 0 | 1 | 0

13. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 78
Description: as for outcome 10
Time Frame: Day 78
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
Participants
  None | 9 | 8 | 8 | 6
  Very mild | 4 | 4 | 5 | 5
  Mild | 0 | 0 | 1 | 0

14. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 92
Description: as for outcome 10
Time Frame: Day 92
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 12 | 14 | 11
Participants
  None | 7 | 7 | 7 | 5
  Very mild | 6 | 5 | 6 | 6
  Mild | 0 | 0 | 1 | 0

15. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 120
Description: as for outcome 10
Time Frame: Day 120
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 13 | 11 | 14 | 11
Participants
  None | 9 | 6 | 6 | 6
  Very mild | 4 | 5 | 6 | 5
  Mild | 0 | 0 | 2 | 0

16. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 162
Description: as for outcome 10
Time Frame: Day 162
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 12 | 11 | 14 | 11
Participants
  None | 9 | 7 | 6 | 7
  Very mild | 3 | 4 | 6 | 4
  Mild | 0 | 0 | 2 | 0

17. Primary Outcome: Number of Participants With Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Score at Day 218
Description: as for outcome 10
Time Frame: Day 218
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 12 | 11 | 14 | 11
Participants
  None | 9 | 7 | 6 | 6
  Very mild | 3 | 4 | 7 | 5
  Mild | 0 | 0 | 1 | 0

18. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline, Day 8, 22, 50, 78 and 92
Population: Per protocol set (PPS) included all participants who were enrolled in the study, received study medication at least once and had at least one efficacy evaluation. Last observation carried forward (LOCF) imputation method was used. Here 'n' signifies participants evaluable for this measure at specified time point for each arm group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Baseline (n = 14, 14, 14, 14) | 61.9 (12.39) | 60.7 (17.28) | 60.4 (16.76) | 63.9 (15.58)
  Day 8 (n = 14, 14, 13, 14) | 60.0 (13.85) | 59.6 (19.44) | 57.8 (17.21) | 62.6 (15.33)
  Day 22 (n = 14, 14, 14, 14) | 56.8 (13.19) | 58.1 (19.59) | 57.1 (16.10) | 60.4 (13.15)
  Day 50 (n = 14, 14, 14, 14) | 57.9 (17.49) | 60.0 (20.47) | 56.5 (15.04) | 62.8 (13.89)
  Day 78 (n = 14, 14, 14, 14) | 56.4 (17.07) | 60.4 (20.05) | 57.2 (18.55) | 59.9 (13.03)
  Day 92 (n = 14, 14, 14, 14) | 56.4 (17.79) | 60.2 (20.38) | 57.4 (17.83) | 60.6 (13.52)

19. Secondary Outcome: Number of Participants With Clinical Global Impression Severity (CGI-S) Score
Description: The CGI-S rating scale is a 7 point (1-absent, 2-minimal, 3-mild, 4-moderate, 5-moderate severe, 6-severe, 7-extreme) global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "normal, not at all ill" and a rating of 7 is equivalent to "among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Day 8, 22, 50, 78 and 92
Population: The PPS included all participants who were enrolled in the study, received study medication at least once and had at least one efficacy evaluation. LOCF imputation method was used. Here 'n' signifies participants evaluable for this measure at specified time point for each arm group.
Measure: Number; unit: Participants
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14
Participants
  Baseline, Minimal (n=14,14,14,14) | 3 | 4 | 3 | 1
  Baseline, Mild (n=14,14,14,14) | 8 | 6 | 10 | 8
  Baseline, Moderate (n=14,14,14,14) | 3 | 3 | 1 | 5
  Baseline, Moderate severe (n=14,14,14,14) | 0 | 1 | 0 | 0
  Day 8, Minimal (n=14,14,13,14) | 3 | 3 | 3 | 1
  Day 8, Mild (n=14,14,13,14) | 8 | 7 | 9 | 10
  Day 8, Moderate (n=14,14,13,14) | 3 | 2 | 1 | 3
  Day 8, Moderate severe (n=14,14,13,14) | 0 | 2 | 0 | 0
  Day 22, Minimal (n=14,14,14,14) | 4 | 5 | 4 | 2
  Day 22, Mild (n=14,14,14,14) | 8 | 5 | 9 | 9
  Day 22, Moderate (n=14,14,14,14) | 2 | 3 | 1 | 3
  Day 22, Moderate severe (n=14,14,14,14) | 0 | 1 | 0 | 0
  Day 50, Minimal (n=14,14,14,14) | 5 | 5 | 3 | 0
  Day 50, Mild (n=14,14,14,14) | 7 | 4 | 10 | 13
  Day 50, Moderate (n=14,14,14,14) | 1 | 3 | 1 | 0
  Day 50, Moderate severe (n=14,14,14,14) | 1 | 2 | 0 | 1
  Day 78, Minimal (n=14,14,14,14) | 6 | 5 | 5 | 1
  Day 78, Mild (n=14,14,14,14) | 6 | 4 | 8 | 12
  Day 78, Moderate (n=14,14,14,14) | 1 | 3 | 0 | 1
  Day 78, Moderate severe (n=14,14,14,14) | 1 | 2 | 1 | 0
  Day 92, Minimal (n=14,14,14,14) | 5 | 4 | 5 | 1
  Day 92, Mild(n=14,14,14,14) | 7 | 5 | 8 | 11
  Day 92, Moderate (n=14,14,14,14) | 1 | 3 | 0 | 2
  Day 92, Moderate severe (n=14,14,14,14) | 1 | 2 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Paliperidone Palmitate 50 mg | Paliperidone Palmitate 100 mg | Paliperidone Palmitate 150 mg | Paliperidone Palmitate 150/ 50 mg
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14 | 2/14 | 3/14
Other Adverse Events (participants affected / at risk) | 14/14 | 14/14 | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone Palmitate 50 mg (N=14) | Paliperidone Palmitate 100 mg (N=14) | Paliperidone Palmitate 150 mg (N=14) | Paliperidone Palmitate 150/ 50 mg (N=14)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neuroleptic malignant syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate 50 mg (N=14) | Paliperidone Palmitate 100 mg (N=14) | Paliperidone Palmitate 150 mg (N=14) | Paliperidone Palmitate 150/ 50 mg (N=14)
Nasopharyngitis (Infections and infestations) | 5 | 4 | 4 | 4
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Purulence (Infections and infestations) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Psychiatric symptom (Psychiatric disorders) | 5 | 6 | 3 | 3
Insomnia (Psychiatric disorders) | 3 | 3 | 4 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 0
Hypochondriasis (Psychiatric disorders) | 0 | 0 | 1 | 1
Abulia (Psychiatric disorders) | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 1 | 2
Akathisia (Nervous system disorders) | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Delayed sleep phase (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 1 | 3 | 2
Injection site erythema (General disorders) | 1 | 1 | 2 | 1
Injection site induration (General disorders) | 2 | 1 | 2 | 0
Thirst (General disorders) | 0 | 2 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Blood prolactin increased (Investigations) | 11 | 9 | 13 | 10
Weight increased (Investigations) | 4 | 2 | 3 | 2
Weight decreased (Investigations) | 3 | 3 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 3
Blood triglycerides increased (Investigations) | 0 | 0 | 2 | 2
White blood cell count increased (Investigations) | 1 | 0 | 2 | 1
Blood prolactin decreased (Investigations) | 1 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1
Blood chloride decreased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0
Blood triglycerides decreased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 1
Urine ketone body present (Investigations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Device breakage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No